CLINICAL TRIAL: NCT05921617
Title: A Cohort Study of Musculoskeletal Health in Patients With Breast Cancer During Aromatase Inhibitors Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Feng Jing, Principal Investigator, Fudan University
Other Study IDs: FJing
Record Dates: First submitted 2023-06-06; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Musculoskeletal Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation group
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Routine care

SUMMARY:
Postmenopausal women with hormone receptor-positive breast cancer are now prescribed aromatase inhibitors with 5 years or longer durations of therapy as recommended by clinical guidelines, which contributes to reducing breast cancer recurrence. However, aromatase inhibitors treatment is associated with a high incidence of musculoskeletal symptoms (MSS), often described as symmetrical pain, soreness in the joints, musculoskeletal pain, and joint stiffness, which even leads to bone loss, osteoporosis, and fractures. MSS reduces patients' quality of life and compliance with aromatase inhibitors therapy in up to one-half of women undergoing adjuvant aromatase inhibitors therapy, potentially compromising breast cancer outcomes. Therefore, this study aimed to monitor the musculoskeletal health of breast cancer patients during endocrine therapy to provide references for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Postoperative early breast cancer；
2. Hormone receptor-positive breast cancer diagnosed by pathology；
3. Aromatase inhibitor therapy (e.g., anastrozole, letrozole, exemestane) was initiated within 3 months;
4. Postmenopausal women, or premenopausal or perimenopausal women taking ovarian function inhibitors;
5. Informed consent and voluntary participation in the study.

Exclusion Criteria:

1. Breast cancer recurrence or distant metastasis;
2. With other malignant tumors;
3. With cognitive or psychiatric disorders.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Study Population: Postoperative patients with hormone receptor-positive breast cancer and treated with aromatase inhibitors in Shanghai Cancer Center, Fudan University, Shanghai, China.
Sampling Method: Non-Probability Sample
Enrollment: 870 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2025-04-27 (Estimated); Study Completion 2025-04-27 (Estimated)

PRIMARY OUTCOMES:
Changes in hand function | Baseline, 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months.
  Measured with score for assessment and quantification of chronic rheumatic affections of the hands (SACRAH).
Changes in wrist function | Baseline, 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months.
  Measured with Boston Carpal Tunnel Questionnaire (BCTQ).
Changes in knee or hip joint function | Baseline, 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months.
  Measured with Western Ontario and McMaster Osteoarthritis Index (WOMAC).

SECONDARY OUTCOMES:
Grip strength | Baseline, 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months.
  Measured with CAMRY EH101 electronic grip strength meter (Made in China).
Bone mineral density | Baseline, 12 months, and 24 months.
  Measured with Lunar iDXA (Made in China).
Depression and Anxiety | Baseline, 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months.
  Measured with the Patient Health Questionnaire for Depression and Anxiety (PHQ-4).
Medication adherence | Baseline, 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months.
  Measured with self-reported medication adherence visual analogue scale (VAS).

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.